CLINICAL TRIAL: NCT01779037
Title: IRF-PAI Functional Outcomes Data(With FIM Instrument Variables)
Status: Terminated | Type: Observational
Sponsor: Uniform Data System for Medical Rehabilitation (Other)
Responsible Party: Sponsor
Other Study IDs: IRFPAIdata
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Heart and Blood Disease; Muscle, Bone and Cartilage Disease; Nervous System Diseases; Skin and Connective Tissue Disease; Wounds and Injuries
MeSH Terms: conditions — Hematologic Diseases; Cartilage Diseases; Nervous System Diseases; Connective Tissue Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inpatient Rehabilitation Patients

SUMMARY:
IRF-PAI Functional Outcomes Data, including FIM instrument variables

DETAILED DESCRIPTION:
United States IRF functional outcomes, medical and socio-demographic data for years 2002-2015

ELIGIBILITY:
Inclusion Criteria:

* Admission to an inpatient rehabilitation facility

Exclusion Criteria:

* Admission to acute, SNF setting, etc.

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: inpatient rehabilitation patients
Sampling Method: Non-Probability Sample
Dates: Start 2001-01; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
IRF-PAI Assessment Instrument(including the FIM instrument) | admission/discharge

CONTACTS AND LOCATIONS:
Locations (1):
- UDSMR, Buffalo, New York, United States

REFERENCES:
- See also: Related Info — http://www.udsmr.org